CLINICAL TRIAL: NCT04444557
Title: Effect of COvid-19 on Mental Health in Syrian and Turkish Maintenance HemoDialysis Patients: COST-HD Study
Acronym: COST-HD
Status: Completed | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Nuri Baris Hasbal, Principal Investigator, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: 200620
Record Dates: First submitted 2020-06-21; First posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Depression; Hemodialysis
Keywords: hemodialysis; depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Turkish hemodialysis patients: Turkish patients undergoing in-center hemodialysis
  Interventions: Other: Beck Depression Inventory (BDI)
- Temporarily protected Syrian hemodialysis patients: Temporarily protected Syrian patients undergoing in-center hemodialysis
  Interventions: Other: Beck Depression Inventory (BDI)

INTERVENTIONS:
Other: Beck Depression Inventory (BDI) — The Beck Depression Inventory (BDI) is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression

SUMMARY:
SARS-COV infection first has begun at Wuhan, China, and then became a pandemic. The first COVID-19 case has been reported on March 11, 2020, in Turkey. People older than 65 years old have been locked down on March 21 and people younger than 20 years old locked down at April 03. A total lockdown has been done a few times lasting for 3 or 4 days, especially at weekends.

Renal replacement modalities have been affected in different ways during the pandemic. Patients with kidney transplantation and patients performing home hemodialysis or peritoneal dialysis have been advised to perform self-isolation at homes. However, center hemodialysis patients continued to come dialysis centers obligatorily.

Syrian civil war has been continuing since 2011, and Turkey has accepted millions of Syrian people in a position called temporary protection. There are many Syrian center hemodialysis patients both in Turkey and in our unit. The investigators do not know if pandemic affected Syrian patients different than Turkish ones. The aim of this study is to compare beck depression scores of Turkish and Syrian patients undergoing hemodialysis during the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old
* Hemodialysis history of more than three months

Exclusion Criteria:

* Patients who can not speak Turkish or Arabic,
* Not volunteer to fill the form
* History of hospitalization for any reason during the pandemic time,
* History of COVID-19 before the questionnaire (Beck Depression Inventory)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing in-center hemodialysis in Sisli Hamidiye Etfal Training and Research hospital (22 patients excluded from the study in accordance with exclusion criteria)
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2020-04-17 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Score of Beck Depression Inventory | through study completion, an average of 6 months
  Total score of Beck Depression Inventory (Minimin score: 0, Maximum score: 63; higher scores mean worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Sevinc, MD, Principal Investigator — Sisli Hamidiye Etfal Training and Research Hospital
Locations (1):
- Sisli Hamidiye Etfal Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
If requested, IPD will be shared